CLINICAL TRIAL: NCT03248414
Title: Investigation of Anti-obesity Properties of Lactobacillus Sakei in Obese Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1511/324-002
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus sakei (Experimental): 2 packs per day
  Interventions: Dietary Supplement: Lactobacillus sakei
- Control (Placebo Comparator): 2 packs per day
  Interventions: Dietary Supplement: Lactobacillus sakei

INTERVENTIONS:
Dietary Supplement: Lactobacillus sakei — 1 pack contained 5 x 109 cfu

SUMMARY:
In this study, we are going to investigate the efficacy of Lactobacillus Sakei on reduction of fat mass assessed by DEXA compared to plaebo.

DETAILED DESCRIPTION:
We are going to enroll subjects whose BMI is equal to higher than 25, and randomly assigned study material or placebo at 1:1 ratio. The treatment duration is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 20-65 years
* BMI equal to higher than 25 kg/m2

Exclusion Criteria:

* under anti-obesity medication
* uncontrolled diabetes
* uncontrolled hypertension
* any medications can influence to body weight such as thiazolidinedione, GLP-1 analogue, SGLT2 inhibitor, diuretics
* thyroid function test abnormality
* malignancy within 5 years
* immune compromised hosts or under immune suppressants
* antibiotics or probiotics withing 2 weeks
* any intervention to reduce body weight within 6 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Fat mass change in 12-week | 12 weeks
  fat mass is measured by DEXA

SECONDARY OUTCOMES:
Changes in body weight | 12 weeks
  body weight change
Changes in waist circumference | 12 weeks
  Waist circumference change
Glucose metabolism | 12 weeks
  Changes in HbA1c
Glucose metabolism | 12 weeks
  Changes in fasting glucose concentration
Glucose metabolism | 12 weeks
  Changes in insulin resistance
Glucose metabolism | 12 weeks
  Changes in beta-cell function

OTHER OUTCOMES:
GI adverse effect | 12 weeks
  incidence of gastrointestinal discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim S, Moon JH, Shin CM, Jeong D, Kim B. Effect of Lactobacillus sakei, a Probiotic Derived from Kimchi, on Body Fat in Koreans with Obesity: A Randomized Controlled Study. Endocrinol Metab (Seoul). 2020 Jun;35(2):425-434. doi: 10.3803/EnM.2020.35.2.425. Epub 2020 Jun 24. PMID 32615727